CLINICAL TRIAL: NCT03676192
Title: A Double-Blind, Randomized, Active-Controlled, Parallel-Group, Phase 3 Study to Compare Efficacy and Safety of CT-P16 and EU-Approved Avastin as First-Line Treatment for Metastatic or Recurrent Non-Squamous Non-Small Cell Lung Cancer
Brief Title: To Compare Efficacy and Safety of CT-P16 and European Union-Approved Avastin as First-Line Treatment for Metastatic or Recurrent Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P16 3.1
Record Dates: First submitted 2018-09-06; First posted 2018-09-18 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Adenocarcinoma of Lung
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P16 (Experimental): Drug: Bevacizumab 15mg/kg IV of CT-P16 will be administered every 3 weeks up to 6 cycles during the Induction Study Period and every 3 weeks until Progressive Disease (PD) or intolerable toxicity during the Maintenance Period.
  Interventions: Drug: CT-P16
- Avastin (Active Comparator): Drug: Bevacizumab 15mg/kg IV of EU-approved Avastin will be administered every 3 weeks up to 6 cycles during the Induction Study Period and every 3 weeks until PD or intolerable toxicity during the Maintenance Period.
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: CT-P16 — 15mg/kg IV of CT-P16 every 3 weeks up to 6 cycles in the induction study period and every 3 weeks until PD occurs in the maintenance study period.
  Arms: CT-P16
Drug: Avastin — 15mg/kg IV of Avastin every 3 weeks up to 6 cycles in the induction study period and every 3 weeks until PD occurs in the maintenance study period.
  Arms: Avastin

SUMMARY:
To demonstrate that CT-P16 is similar to EU-Approved Avastin in terms of efficacy as determined by objective response rate (ORR) during the Induction Study Period

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as recurrent disease or stage IV
* has at least 1 measurable lesion by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1

Exclusion Criteria:

* has predominantly squamous cell histology non-small cell lung cancer
* had surgery for metastatic non-squamous non-small cell lung cancer (nsNSCLC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Andric Z, Moiseenko F, Makharadze T, Oleksiienko A, Yanez Ruiz E, Kim S, Ahn K, Park T, Ju H, Baek EH, Kwon S, Chang I, Kim S, Kim H, Lee E, Verschraegen C. Long-term results of a randomized controlled trial of biosimilar CT-P16 and reference bevacizumab in patients with metastatic or recurrent non-small cell lung cancer. Cancer Treat Res Commun. 2025;44:100970. doi: 10.1016/j.ctarc.2025.100970. Epub 2025 Jul 24. PMID 40795416
- [Derived] Verschraegen C, Andric Z, Moiseenko F, Makharadze T, Shevnya S, Oleksiienko A, Yanez Ruiz E, Kim S, Ahn K, Park T, Park S, Ju H, Ohe Y. Candidate Bevacizumab Biosimilar CT-P16 versus European Union Reference Bevacizumab in Patients with Metastatic or Recurrent Non-Small Cell Lung Cancer: A Randomized Controlled Trial. BioDrugs. 2022 Nov;36(6):749-760. doi: 10.1007/s40259-022-00552-8. Epub 2022 Sep 28. PMID 36169807

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin: Drug: Bevacizumab 15mg/kg IV of European Union (EU)-approved Avastin will be administered every 3 weeks up to 6 cycles during the Induction Study Period and every 3 weeks until Progressive Disease (PD) or intolerable toxicity during the Maintenance Period.
  Avastin: 15mg/kg IV of Avastin every 3 weeks up to 6 cycles in the induction study period and every 3 weeks until PD occurs in the maintenance study period.
- CT-P16: Drug: Bevacizumab 15mg/kg IV of CT-P16 will be administered every 3 weeks up to 6 cycles during the Induction Study Period and every 3 weeks until PD or intolerable toxicity during the Maintenance Period.
  CT-P16: 15mg/kg IV of CT-P16 every 3 weeks up to 6 cycles in the induction study period and every 3 weeks until PD occurs in the maintenance study period.
Period: Induction Study Period
Arm/Group | Avastin | CT-P16
Started | 347 | 342
Completed | 241 | 258
Not Completed | 106 | 84
Not completed — Adverse Event | 21 | 20
Not completed — Death | 23 | 20
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 6 | 3
Not completed — Progressive Disease | 32 | 21
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 20 | 15
Period: Maintenance Study Period
Arm/Group | Avastin | CT-P16
Started (The number of patients who started Maintenance Study Period is not equal to the number who completed Induction Study Period.) | 227 | 239
Completed (Patients received the study drug until progressive disease, interolerable toxicity, or end of study, whichever occured first.) | 227 | 239
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population: All randomized patients who were randomly assigned to study drug regardless of whether or not any study treatment dosing was completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P16 | Avastin | Total
Number analyzed (Participants) | 342 | 347 | 689
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.01) | 61.5 (9.42) | 61.4 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 125 | 244
  Male | 223 | 222 | 445
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 9 | 18
  Asian | 59 | 55 | 114
  Black or African American | 2 | 1 | 3
  White or Caucasian | 264 | 264 | 528
  Other | 8 | 18 | 26
Disease Status [Count of Participants; unit: Participants]
  Recurrent | 25 | 33 | 58
  Metastatic | 317 | 314 | 631
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, but ambulatory and able to carry out work of light nature or sedentary nature; 2 = Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0 | 105 | 110 | 215
    Grade 1 | 237 | 237 | 474

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) During the Induction Study Period From Central Review
Description: The ORR was defined as the proportion of patients with a confirmed Best Overall Response (BOR) of CR or PR (the 'responder'). All other patients except responders were considered as non-responders, including patients without post-baseline tumor assessment.
Time Frame: Induction Study Period (around 18 weeks)
Population: Intent-to-Treat (ITT) population: All randomized patients who were randomly assigned to study drug regardless of whether or not any study treatment dosing was completed.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 342 | 347
percentage of responders | 42.40 [37.16 to 47.64] | 42.07 [36.88 to 47.27]
Statistical Analysis 1: Comparison: CT-P16 vs Avastin; Logistic regression model including treatment groups (CT-P16 and EU-approved Avastin) as a fixed effect and region (EMEA vs. America vs. Asia), sex (female vs. male), disease status at baseline (recurrence vs. metastatic), and ECOG performance score at baseline (0 vs. 1) as covariates was used; Test type: Equivalence — The similarity criterion had been set such that the confidence limits of the 95% confidence interval (CI) of the difference of ORR from each treatment group was entirely bounded by the interval (-12.5, 12.5); Risk Difference (RD) = 0.40, 95% CI 2-sided [-7.02 to 7.83]
Statistical Analysis 2: Comparison: CT-P16 vs Avastin; Log-binomial regression model including treatment groups (CT-P16 and EU-approved Avastin) as a fixed effect and region (EMEA vs. America vs. Asia), sex (female vs. male), disease status at baseline (recurrence vs. metastatic), and ECOG performance score at baseline (0 vs. 1) as covariates was used; Test type: Equivalence — The similarity criterion had been set such that the confidence limits of the 90% confidence interval (CI) of the ratio of ORR from each treatment group was entirely bounded by the interval (0.7368, 1.3572); Risk Ratio (RR) = 1.0136, 90% CI 2-sided [0.8767 to 1.1719]

2. Secondary Outcome: Response Duration From Central Review
Description: Response duration was defined as time between initial response (CR or PR) that is confirmed by the subsequent assessment after study treatment administration and PD/recurrence or death from any cause, whichever occurs first.
Time Frame: Tumor assessments were assessed every 2 cycles during the Induction Study Period, every 3 cycles during the Maintenance Study Period, and at the EOT visit. The median follow-up time from randomization was 12.86 months.
Population: Patients who have confirmed BOR of CR or PR from ITT population (All randomized patients who were randomly assigned to study drug regardless of whether or not any study treatment dosing was completed).
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 156 | 160
Proportion of participants
  6 months | 0.60 [0.51 to 0.67] | 0.56 [0.48 to 0.64]
  12 months | 0.17 [0.11 to 0.25] | 0.25 [0.18 to 0.32]
  24 months | 0.09 [0.04 to 0.15] | 0.10 [0.06 to 0.17]
  36 months | 0.08 [0.04 to 0.14] | 0.06 [0.02 to 0.12]

3. Secondary Outcome: Time to Progression From Central Review
Description: Time to progression was defined as time from randomization to determined PD/recurrence.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 342 | 347
Proportion of participants
  6 months | 0.83 [0.78 to 0.87] | 0.81 [0.76 to 0.85]
  12 months | 0.29 [0.23 to 0.35] | 0.34 [0.27 to 0.40]
  24 months | 0.11 [0.07 to 0.17] | 0.11 [0.07 to 0.16]
  36 months | 0.10 [0.06 to 0.16] | 0.06 [0.03 to 0.12]

4. Secondary Outcome: Progression Free Survival From Central Review
Description: Progression-free survival was defined as time from randomization to determined PD/recurrence or death from any cause, whichever occurs first.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 342 | 347
Proportion of participants
  6 months | 0.73 [0.68 to 0.78] | 0.71 [0.66 to 0.76]
  12 months | 0.23 [0.19 to 0.29] | 0.28 [0.23 to 0.34]
  24 months | 0.08 [0.05 to 0.12] | 0.09 [0.06 to 0.13]
  36 months | 0.06 [0.03 to 0.10] | 0.04 [0.02 to 0.08]
Statistical Analysis 1: Comparison: CT-P16 vs Avastin; Adjusted stratified Cox regression model is used to estimate the hazard ratio and its 95% CI for receiving CT-P16 compared with receiving EU-approved Avastin using region (EMEA vs. America vs. Asia), sex (female vs. male), disease status at baseline (recurrence vs. metastatic), and ECOG performance score at baseline (0 vs. 1) as stratification factors; Test type: Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.10]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from randomization to death from any cause.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 342 | 347
Proportion of participants
  12 months | 0.66 [0.60 to 0.71] | 0.62 [0.56 to 0.67]
  24 months | 0.35 [0.29 to 0.40] | 0.34 [0.29 to 0.40]
  36 months | 0.19 [0.14 to 0.24] | 0.21 [0.16 to 0.26]
Statistical Analysis 1: Comparison: CT-P16 vs Avastin; [analysis description as in outcome 4, analysis 1]; Test type: Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.77 to 1.19]

6. Secondary Outcome: Trough Serum Concentrations During the Induction Study Period
Description: Pharmacokinetic samples were collected on Day 1 of each cycle (prior to the beginning of the study drug administration) in the Induction Study Period.
Time Frame: Induction Study Period. Pharmacokinetic samples were collected on Day 1 of each cycle in Induction Study Period.
Population: Pharmacokinetic (PK) population: all randomly assigned patients who received at least 1 full dose of study drug (CT-P16 or Avastin) and who had at least 1 post-treatment PK result. Patients who received incorrect treatment during the Induction Study Period were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 327 | 323
μg/L
  Induction Cycle 1: number analyzed (Participants) | 318 | 316
  Induction Cycle 1 | 50426.3 (39847.34) | 52515.7 (32356.13)
  Induction Cycle 2: number analyzed (Participants) | 302 | 287
  Induction Cycle 2 | 73127.7 (35883.59) | 81533.7 (52567.34)
  Induction Cycle 3: number analyzed (Participants) | 283 | 269
  Induction Cycle 3 | 93100.6 (50495.29) | 95878.8 (53977.69)
  Induction Cycle 4: number analyzed (Participants) | 268 | 254
  Induction Cycle 4 | 96445.2 (45597.95) | 101583.1 (46275.62)
  Induction Cycle 5: number analyzed (Participants) | 252 | 238
  Induction Cycle 5 | 108957.3 (55135.16) | 108512.5 (49823.61)
  Induction Cycle 6: number analyzed (Participants) | 246 | 228
  Induction Cycle 6 | 116188.2 (58735.47) | 114849.6 (56309.70)

7. Secondary Outcome: Patients With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (NAb) at Anytime During the Whole Study Period
Description: Immunogenicity was assessed on Day 1 of Cycle 1 (pre-dose), every 2 cycles during the Induction Study Period, and every 3 cycles during the Maintenance Study Period and End of Treatment (EOT) visit. In the Follow-Up Period, immunogenicity was assessed once at the first visit of the Follow-Up Period (ninth week).
Time Frame: Immunogenicity was assessed Day 1 of Cycle 1 (predose), every 2 cycles during the Induction Study Period, every 3 cycles during the Maintenance Study Period, EOT visit, and at the first visit of Follow-up period.
Population: Safety Population: all randomly assigned patients who received at least 1 dose (partial or full) of study drug (CT-P16 or Avastin). Patients receiving at least 1 dose of CT-P16 at any time of during the treatment period were analyzed under the CT-P16 treatment group. Three patients who were randomized to Avastin treatment group were analyzed under the CT-P16 treatment group since the patients incorrectly received CT-P16 during the treatment period.
Measure: Number; unit: participants
Arm/Group | CT-P16 | Avastin
Number analyzed (Participants) | 345 | 344
participants
  Subject with at least 1 positive ADA result after the first infusion | 81 | 90
  Patients with at least 1 positive NAb result after the first infusion | 12 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the informed consent form is signed until up to 28 days from last dose of study drug, regardless of the relationship to the study drug, regardless of the relationship to the study drug.
Description: Three patients who were randomized to Avastin treatment group were analyzed under the CT-P16 treatment group since the patients incorrectly received CT-P16 during the treatment period.
Arm/Group | CT-P16 | Avastin
All-Cause Mortality (participants affected / at risk) | 24/345 | 25/344
Serious Adverse Events (participants affected / at risk) | 69/345 | 73/344
Other Adverse Events (participants affected / at risk) | 332/345 | 320/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P16 (N=345) | Avastin (N=344)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Food Poisoning (Gastrointestinal disorders) | 2 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatic Pseudocyst Rupture (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 2 | 3
Fatigue (General disorders) | 0 | 1
Hyperthermia Malignant (General disorders) | 1 | 0
Sudden Death (General disorders) | 2 | 3
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Anaphylactic Shock (Immune system disorders) | 1 | 0
Contrast Media Reaction (Immune system disorders) | 1 | 0
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
COVID-19 Pneumonia (Infections and infestations) | 5 | 4
Infectious Pleural Effusion (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 9 | 10
Pneumonia Mycoplasmal (Infections and infestations) | 0 | 1
Renal Abscess (Infections and infestations) | 1 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic Shock (Infections and infestations) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 2
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Laryngeal Nerve Dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Neurological Symptom (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 0 | 1
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Renal Infarct (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oesophagobronchial Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Accelerated Hypertension (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 3 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P16 (N=345) | Avastin (N=344)
Anaemia (Blood and lymphatic system disorders) | 109 | 93
Leukopenia (Blood and lymphatic system disorders) | 30 | 23
Neutropenia (Blood and lymphatic system disorders) | 75 | 55
Thrombocytopenia (Blood and lymphatic system disorders) | 63 | 48
Constipation (Gastrointestinal disorders) | 38 | 33
Diarrhoea (Gastrointestinal disorders) | 43 | 47
Nausea (Gastrointestinal disorders) | 74 | 65
Vomiting (Gastrointestinal disorders) | 30 | 30
Asthenia (General disorders) | 63 | 54
Fatigue (General disorders) | 45 | 40
Pyrexia (General disorders) | 22 | 17
Pneumonia (Infections and infestations) | 15 | 18
Urinary Tract Infection (Infections and infestations) | 20 | 9
Alanine Aminotransferase Increased (Investigations) | 24 | 19
Aspartate Aminotransferase Increased (Investigations) | 23 | 17
Gamma-Glutamyltransferase Increased (Investigations) | 22 | 19
Neutrophil Count Decreased (Investigations) | 16 | 19
Platelet Count Decreased (Investigations) | 29 | 23
Weight Decreased (Investigations) | 34 | 31
Decreased Appetite (Metabolism and nutrition disorders) | 43 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 18
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 18 | 20
Headache (Nervous system disorders) | 25 | 21
Neuropathy Peripheral (Nervous system disorders) | 53 | 50
Paraesthesia (Nervous system disorders) | 35 | 29
Peripheral Sensory Neuropathy (Nervous system disorders) | 35 | 35
Proteinuria (Renal and urinary disorders) | 44 | 44
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 220 | 218
Hypertension (Vascular disorders) | 36 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03676192/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT03676192/SAP_001.pdf